CLINICAL TRIAL: NCT04623476
Title: PAtophysiological, Nodal-based Approach for Crohn's Disease Excision: A PILOT Study
Brief Title: PAtophysiological, Nodal-based Approach for Crohn's Disease Excision
Acronym: PANACEAPILOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Associate Professor, Head of Department, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112/20
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Crohn Disease; Crohn's Ileocolitis
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Prospective pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pathophysiological Excision for Chron's disease (Experimental): Consecutive patients (>18 years old) with a surgical indication for ileocolic Crohn's disease, at their first operation for CD
  Interventions: Procedure: Pathophysiological Excision for Crohn's disease

INTERVENTIONS:
Procedure: Pathophysiological Excision for Crohn's disease — Pathophysiological excision for Crohn's (PEC) requires a medio-lateral approach and a high vascular tie, which enables excision of lymph nodes draining the disease bowel. This procedure should not alter length of bowel resection and no additional risks are foreseen. A latero-lateral anastomosis will be fashioned following current guidelines.
  Other Names: PEC

SUMMARY:
Single centre prospective pilot study on surgery for Crohn's disease (CD). CD universally recurs after surgery and no technique so far has been proven to reduce recurrence.

The investigators speculate that a different surgical technique, based on pathophysiology of the disease may prove successful in reducing rates of recurrence.

Consecutive CD patients with a surgical indication for ileocolic disease will receive an extended procedure including a lymphadenectomy (Pathophysiologic excision for Crohn's disease).

Primary outcome will be endoscopic recurrence rates at 6 and 12 months from surgery.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing surgery for ileocaecal/ileocolic CD in the Minimally Invasive Unit at Policlinico Tor Vergata are eligible to be enrolled.
* Informed consent

Exclusion Criteria:

* Crohn's Disease with a different localisation
* Recurrent disease
* Extensive jejunitis
* <18 years of age
* Cancer as primary indication for surgery
* Followed by gastroenterologists outside our centre, due to loss of follow up
* Ileostomy. If a patient undergoes ileostomy fashioning he will be excluded from the study and this will be reported

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of endoscopic CD recurrence | 6 months
  Endoscopic Rutgeerts score >1
Rate of endoscopic CD recurrence | 12 months
  Endoscopic Rutgeerts score >1

SECONDARY OUTCOMES:
Rate of overall postoperative complications | 30 days
  Clavien Dindo I-V
Rate of major postoperative complications | 30 days
  Clavien Dindo III-V
Overall and Disease specific Quality of life | 6 months
  Inflammatory Bowel Disease Questionnaire (32 to 224 with higher scores representing better quality of life)
Overall and Disease specific Quality of life | 6 months
  Inflammatory Bowel Disease-Control (Q 1-3 with higher scores representing better quality of life)
Overall and Disease specific Quality of life | 6 months
  Cleveland Global Quality of Life score (0-1 with with higher scores representing better quality of life)
Overall and Disease specific Quality of life | 12 months
  Inflammatory Bowel Disease Questionnaire (32 to 224 with higher scores representing better quality of life)
Overall and Disease specific Quality of life | 12 months
  Inflammatory Bowel Disease-Control Q1-3 (0-18 with higher scores representing better quality of life)
Overall and Disease specific Quality of life | 12 months
  Cleveland Global Quality of Life score (0-1 with higher scores representing better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe S Sica, MD, PhD, Principal Investigator — Università di Roma Tor Vergata
Locations (1):
- Policlinico Tor Vergata, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No